CLINICAL TRIAL: NCT07267104
Title: SAGE-NIV: Surveillance and Artificial Intelligence Guidance for Exacerbations in COPD Patients With Home Non-Invasive Ventilation
Brief Title: Mathematical Analysis of Signals and Clinical Parameters Provided by Non-invasive Home Ventilation Devices
Acronym: SAGE-NIV
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Cristina Lalmolda-Puyol, NIV coordinator Neumology Service, Corporacion Parc Tauli
Other Study IDs: SAGE-NIV; SEPAR PII-NIV (Other Grant/Funding Number: Sociedad española de neumología y cirugía torácica)
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Artificial Intelligent; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study cohort with COPD and NIV patients for at least 6 months: 1. Inclusion criteria:
     * Age between 40 and 80 years.
     * COPD diagnosed by pulmonary function tests.
     * Home NIV therapy with good adherence (minimum daily compliance > 5 hours) for at least 6 months.
     * Users of the ResMed LUMIS 150 ventilator. This is due to the presence of the decoding tool and a larger storage capacity (more than 100 nights) in the removable device of the ventilator.
     * Acute exacerbation requiring hospital admission or home care.
  2. Exclusion criteria:
     * Lack of informed consent.
     * Previous clinical instability defined by the need for antibiotics and/or systemic corticosteroids in the two months prior to the inclusion exacerbation, excluding the 48 hours prior to admission, as this was considered part of the inclusion clinical picture.
  Ethical aspects:
  Patients will receive written information about the study and will also receive verbal explanations to clarify any doubts. Participation is voluntary and the patient may withdraw from the study at any time. No inv
  Interventions: Other: The intervention involves download data of ventilator with clinical dates of the patient and model ventilator and parameters in acute exacebartion fo COPD

INTERVENTIONS:
Other: The intervention involves download data of ventilator with clinical dates of the patient and model ventilator and parameters in acute exacebartion fo COPD — Recruitment:
  * Collection of the clinical variables described in the previous section.
  * Download the data from the commercial ventilator mentioned in the 'Inclusion criteria' section. By default, the option 'all available detailed data' is selected in the menu corresponding to the built-in software.
  * Contact the coordinating centre to obtain an internal study code.
  * Send the contents of the folder corresponding to the recruited patient to the coordinating centre (using an encrypted system).
  Treatment and handling of data:
  * The clinical data collected after anonymisation will be stored on-line using the RedCap platform (https://www.project-redcap.org/). Data downloaded from the ventilator will be identified by a random code and stored on the encrypted Proton platform (https://proton.me/es-es) or similar.
  * Built-in software data:
  Once the file has been received, the 10 days prior to the admission, which will be the reason for recruitment

SUMMARY:
This study will look at people with COPD who use a home breathing machine called non-invasive ventilation (NIV). NIV machines collect information about your breathing, such as air flow, pressure, and mask leaks.

Researchers want to use a computer program, called artificial intelligence (AI), to study this information. The goal is to find early signs that your breathing may be getting worse.

People with COPD who already use NIV at home may join this study. The study does not change your treatment. It only uses the breathing data already recorded by your NIV machine.

The computer program will look for patterns in the data. These patterns may help doctors:

Notice early warning signs of a COPD flare-up Find problems with how you and the machine work together Improve the way NIV is monitored at home The main goal is to create a tool that helps patients and doctors manage home NIV more easily and more safely.

DETAILED DESCRIPTION:
This study proposes the development of an artificial intelligence (AI) system to monitor and analyse detailed non-invasive mechanical ventilation (NIV) data in COPD patients, with the aim of predicting clinical exacerbations and improving home management.

Analysis of data from home NIV devices allows assessment of patient compliance, detection of leaks and asynchronies, and monitoring of upper airway events. However, the potential of these data to improve ventilation management in COPD patients has been limited, in part due to the lack of tools to process and interpret the detailed records. Transforming these data into an open format opens up the possibility of applying artificial intelligence to analyse large amounts of information and develop predictive models.

The multi-centre, observational, longitudinal study design will include COPD patients on NIV therapy who meet adherence criteria. Detailed leak, pressure and flow time data, previously decrypted and converted into a data format readable by analysis software, will be analysed. The identified metrics will be evaluated by machine learning algorithms using techniques such as random forest and neural networks.

Expected outcomes include the development of an automated predictive model to enable early detection of exacerbations and improved patient-ventilator synchronisation, moving towards more efficient and personalised telemonitoring in home NIV management.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years.
* COPD diagnosed by pulmonary function tests.
* Home NIV therapy with good adherence (minimum daily compliance > 5 hours) for at least 6 months.
* Users of the ResMed LUMIS 150 ventilator. This is due to the presence of the decoding tool and a larger storage capacity (more than 100 nights) in the removable device of the ventilator.
* Acute exacerbation requiring hospital admission or home care.

Exclusion Criteria:

* Lack of informed consent.
* Previous clinical instability defined by the need for antibiotics and/or systemic corticosteroids in the two months prior to the inclusion exacerbation, excluding the 48 hours prior to admission, as this was considered part of the inclusion clinical picture.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD with chronic NIV in acute exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean expiratory constant time (seconds) | the 10 days prior to the admission, which will be the reason for recruitment, and the 10 days that will act as a control
  Mean expiratory constant time based on signal reconstruction and development of metrics basics on the data of traces of the patient ventilator detailed registered. They are converted to an open format using the tool provided and then uploaded to the protected data cloud. Signal reconstruction: based on the matrix , a programme has already been developed in Matlab® to reconstruct the signal from the built-in software. The events (arrows) are exactly the same in the built-in software and in the metrics development program. Three channels are imported: leakage, pressure and flow. Individual metrics For the expiratory part, peak expiratory, distance to peak expiratory, time constant, trend changes (points with first derivative = 0), etc. All mathematical development is implemented in in Matlab to facilitate automation.

SECONDARY OUTCOMES:
Mean respiratory rate (RR) rpm | 10 days prior to the admission, which will be the reason for recruitment, and the 10 days that will act as a control
  RR based on the same signal reconstruction based on the matrix with a programme has already been developed in Matlab® to reconstruct the signal from the built-in software ventilator Some of the metrics to be defined are: for inspiration, peak flow, distance to peak flow, number of peaks, inspiratory time constant, etc. For the expiratory part, peak expiratory, distance to peak expiratory, time constant, trend changes (points with first derivative = 0), etc. All mathematical development is implemented in Matlab to facilitate automation.
Mean inspiratory time (seconds) | the 10 days prior to the admission, which will be the reason for recruitment, and the 10 days that will act as a control
  Mean inspiratory time (seconds) obtained by the same signal reconstruction. based on the same signal reconstruction based on the matrix with a programme has already been developed in Matlab® to reconstruct the signal from the built-in software ventilator Some of the metrics to be defined are: for inspiration, peak flow, distance to peak flow, number of peaks, inspiratory time constant, etc. For the expiratory part, peak expiratory, distance to peak expiratory, time constant, trend changes (points with first derivative = 0), etc. All mathematical development is implemented in Matlab to facilitate automation.
Mean Inspiratory time/ total time (s) | 10 days prior to the admission, which will be the reason for recruitment, and the 10 days that will act as a control
  Mean of this realtion based on the same signal reconstruction based on the matrix with a programme has already been developed in Matlab® to reconstruct the signal from the built-in software ventilator Some of the metrics to be defined are: for inspiration, peak flow, distance to peak flow, number of peaks, inspiratory time constant, etc. For the expiratory part, peak expiratory, distance to peak expiratory, time constant, trend changes (points with first derivative = 0), etc. All mathematical development is implemented in Matlab to facilitate automation.
exacerbation previous year (n) | Baseline
  Specified if the patient had an exacerbation or more the previous year, review of clinical history form previous year
FEV1 (%) | Baseline
  FEV1 (%), of the last spirometry, last spirometry previous acute exacerbation
FVC % | Baseline
  FVC% of last spirometry, FVC% of last spirometry previous of acute exacerbation
FEV1/FVC % | Baseline
  FEV1/FVC % OF LAST SPIROMETRY, previous of acute exacerbation
Date of exacerbation (dd/mm/yyyy) | Baseline
  date of admission
Age (years) | Baseline
  age in the admission
Gender (male / female) | Baseline
  gender of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Corporation Parc Tauli de Sabadell, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Redcap and drive account
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Available since 2025, March to December 2026
Access Criteria: Each PI of every center involve in the project